CLINICAL TRIAL: NCT01136512
Title: Metformin Use and Vitamin B12 Deficiency
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 07040
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Vitamin B12 Deficiency; Type 2 Diabetes Mellitus
Keywords: metformin; vitamin B12; type 2 diabetes; methylmalonic acid; deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- metformin use: Patients with type 2 diabetes treated with metformin
- no metformin use: Patients with type 2 diabetes who are not being treated with metformin

SUMMARY:
The primary objective is to determine the incidence of Vitamin B12 deficiency in patients on metformin therapy for diabetes.

ELIGIBILITY:
Inclusion Criteria:Age 20-80; diagnosed with type 2 diabetes for at least 30 days

Exclusion Criteria:known vitamin B12 or folate deficiency; pernicious anemia; on vitamin B12 therapy; hematological malignancy; methotrexate use; alcohol intake greater than two drinks per day; vegetarian diet; previous gastric surgery; inflammatory bowel disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient and hospitalized patients with type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Vitamin B12 level | Single point

SECONDARY OUTCOMES:
methylmalonic acid | single point

CONTACTS AND LOCATIONS:
Overall Officials: Neil Cohen, M.D., Principal Investigator — Staten Island University Hospital
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States